CLINICAL TRIAL: NCT01099501
Title: Oxepa in Multiple Trauma: Prospective, Randomized, Comparative, Double-blind, Controlled Clinical Study
Brief Title: Oxepa in Multiple Trauma
Acronym: OMT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Israeli Ministry of Security (Unknown)
Responsible Party: Principal Investigator, Pierre singer, Professor, MD, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PHMD- OT- 01
Record Dates: First submitted 2010-04-01; First posted 2010-04-07 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-10

CONDITIONS: Multiple Trauma; Head Trauma
Keywords: Mechanical Ventilation
MeSH Terms: conditions — Multiple Trauma; Craniocerebral Trauma | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxepa (Active Comparator): Oxepa (enteral nutrition formula, ABBOTT)will be administered at a dose determined by a patient's energy expenditure and tolerance of enteral feeding.
  Interventions: Dietary Supplement: Oxepa (enteral nutrition formula, ABBOTT), at a dose determined by a patient's energy expenditure and tolerance of enteral feeding.; Dietary Supplement: oxepa
- Control group (Active Comparator): Pulmocare or Jevity (enteral nutrition formula, ABBOTT)will be administered at a dose determined by a patient's energy expenditure and tolerance of enteral feeding.
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Oxepa (enteral nutrition formula, ABBOTT), at a dose determined by a patient's energy expenditure and tolerance of enteral feeding. — Oxepa will be administered(enteral nutrition formula, ABBOTT), at a dose determined by a patient's energy expenditure and tolerance of enteral feeding
  Arms: Oxepa
Dietary Supplement: oxepa — A dose determined by a patient's energy expenditure and tolerance of enteral feeding.
  Arms: Oxepa
Dietary Supplement: Control group — Pulmocare or Jevity (enteral nutrition formula, ABBOTT)will be administered at a dose determined by a patient's energy expenditure and tolerance of enteral feeding.
  Arms: Control group

SUMMARY:
This is a single-center, prospective, randomized, comparative, double-blind controlled clinical study mend to assess the effect of enteral feeding with Oxepa (a fish oil-based nutrition), compared to an isocaloric control, on oxygenation and clinical outcomes in mechanically ventilated trauma patients.

The study population will be adults admitted to the ICU due to multiple-trauma or head trauma as a result of a gun shut, motor vehicle accidents, fall, workplace accident etc.

DETAILED DESCRIPTION:
Primary outcome:

Improvement in oxygenation

Secondary outcomes:

Significant improvement in other clinical and laboratory end points.

Primary endpoint:

Pulmonary function:

Oxygenation (PO2- FIO2 ratio)

* Incidence of ALI
* Length of Ventilation (LOV)

Secondary endpoints:

Rate of complications:

-New organ failure.

Rate of new infections:

-wound infection, bacteremia, ventilation associated pneumonia.

Pain:

-Pain score and analgesic use

Morbidity/ mortality:

* Length of ICU stay
* Length of hospitalization
* 28 day mortality
* Hospital mortality

All patients will commence enteral feeding via a nasogastric or orogastric tube; allocation to either Oxepa or Pulmocare/Jevity (control group) will be determined by randomization code. Patients will be prescribed to receive a daily amount of enteral formula that provides at least 80% of their energy; the latter will be calculated every 48 to 72 hours by Indirect Calorimetric (IC) measurement of Resting Energy Expenditure (REE). Tolerance of EN will be assessed by measurement of Gastric Residual Volume (GRV) every 8 hrs and the mode of feeding will be modified accordingly.

Treatment:

Enrolled patients will be randomly divided into a control group and an intervention group.

Control group treatment:

Will be administered Pulmocare or Jevity (enteral nutrition formula, ABBOTT), at a dose determined by a patient's energy expenditure and tolerance of enteral feeding.

Intervention group treatment:

Will be administered with Oxepa (enteral nutrition formula, ABBOTT), at a dose determined by a patient's energy expenditure and tolerance of enteral feeding.

Treatment duration:

The above formulas will be/delivered until the first of the following occurs:

* patients resume regular oral feeding
* day 28/ discharge from ICU/ exitus
* Patients transferred to Total Parenteral Nutrition Note: the attending physician according to the patient's needs will determine feeding of patients from there on.

Study termination (end of all study procedures):

* day 28/ discharge from ICU
* Patients transferred to Total Parenteral Nutrition before day 3 of the study

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18-90 years with multiple-trauma or head trauma admitted to the ICU.
2. Enteral nutrition can be initiated within 36 hours of admission/ injury.
3. Mechanical ventilation.

Exclusion criteria:

1. Severe underlying systemic disease and /or treatment with immunosuppressive agents.
2. Contra-indication for Enteral Nutrition (mechanical or functional bowel. obstruction, high-output fistula, severe necrotizing pancreatitis).
3. 2nd /3rd degree burns covering > 66% BSA.
4. Pregnancy.
5. Participants under the age of 18.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-04; Primary Completion 2014-05 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Oxygenation (PO2/FIO2 ratio) | 2 years
  PO2/FIO2 ratio; assessed by measuring arterial blood gases (AVL Omni Technology, Graz, Austria) and ventilator settings (10)

SECONDARY OUTCOMES:
TNF-α, CRP (markers of inflammatory response) | 2 years
  Concentration of circulating inflammatory markers: TNF-α, CRP concentrations
Fatty acid composition of RBC phospholipids, including n-3:n-6 ratio (markers of n-3 PUFA incorporation into blood cell membranes) | 2 years
  Fatty acid composition of RBC membrane (thin liquid chromatography)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Singer, MD, Professor, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Campus Beilinson, Petah Tikva, Israel

REFERENCES:
- [Background] MacCallum NS, Evans TW. Epidemiology of acute lung injury. Curr Opin Crit Care. 2005 Feb;11(1):43-9. doi: 10.1097/00075198-200502000-00007. PMID 15659944
- [Background] Bernard GR, Artigas A, Brigham KL, Carlet J, Falke K, Hudson L, Lamy M, Legall JR, Morris A, Spragg R. The American-European Consensus Conference on ARDS. Definitions, mechanisms, relevant outcomes, and clinical trial coordination. Am J Respir Crit Care Med. 1994 Mar;149(3 Pt 1):818-24. doi: 10.1164/ajrccm.149.3.7509706.
- [Background] Moore FA, Moore EE, Jones TN, McCroskey BL, Peterson VM. TEN versus TPN following major abdominal trauma--reduced septic morbidity. J Trauma. 1989 Jul;29(7):916-22; discussion 922-3. doi: 10.1097/00005373-198907000-00003. PMID 2501509
- [Background] Kudsk KA, Croce MA, Fabian TC, Minard G, Tolley EA, Poret HA, Kuhl MR, Brown RO. Enteral versus parenteral feeding. Effects on septic morbidity after blunt and penetrating abdominal trauma. Ann Surg. 1992 May;215(5):503-11; discussion 511-3. doi: 10.1097/00000658-199205000-00013. PMID 1616387
- [Background] Kudsk KA, Minard G, Croce MA, Brown RO, Lowrey TS, Pritchard FE, Dickerson RN, Fabian TC. A randomized trial of isonitrogenous enteral diets after severe trauma. An immune-enhancing diet reduces septic complications. Ann Surg. 1996 Oct;224(4):531-40; discussion 540-3. doi: 10.1097/00000658-199610000-00011. PMID 8857857
- [Background] Moore FA, Moore EE, Kudsk KA, Brown RO, Bower RH, Koruda MJ, Baker CC, Barbul A. Clinical benefits of an immune-enhancing diet for early postinjury enteral feeding. J Trauma. 1994 Oct;37(4):607-15. doi: 10.1097/00005373-199410000-00014. PMID 7932892
- [Background] Todd SR, Gonzalez EA, Turner K, Kozar RA. Update on postinjury nutrition. Curr Opin Crit Care. 2008 Dec;14(6):690-5. doi: 10.1097/MCC.0b013e3283196562. PMID 19005311
- [Background] Singer P, Theilla M, Fisher H, Gibstein L, Grozovski E, Cohen J. Benefit of an enteral diet enriched with eicosapentaenoic acid and gamma-linolenic acid in ventilated patients with acute lung injury. Crit Care Med. 2006 Apr;34(4):1033-8. doi: 10.1097/01.CCM.0000206111.23629.0A. PMID 16484911
- [Background] Green P, Hermesh H, Monselise A, Marom S, Presburger G, Weizman A. Red cell membrane omega-3 fatty acids are decreased in nondepressed patients with social anxiety disorder. Eur Neuropsychopharmacol. 2006 Feb;16(2):107-13. doi: 10.1016/j.euroneuro.2005.07.005. Epub 2005 Oct 21. PMID 16243493
- [Result] Giannoudis PV. Current concepts of the inflammatory response after major trauma: an update. Injury. 2003 Jun;34(6):397-404. doi: 10.1016/s0020-1383(02)00416-3. PMID 12767787
- [Result] Leaver SK, Evans TW. Acute respiratory distress syndrome. BMJ. 2007 Aug 25;335(7616):389-94. doi: 10.1136/bmj.39293.624699.AD. No abstract available. PMID 17717368
- [Result] Singer P, Cohen J: Indirect calorimetry and metabolic monitoring. In Fink M, Abraham E (eds), Textbook of Critical Care, Springer eds (Berlin), 2005 pp.]
- [Result] Gaynes RP, Horan TC. Surveillance of Nosocomial Infections.In: Mayhall CG, editor. Hospital Epidemiology and Infection Control. Philadelphia: Lippincott Williams & Wilkins,1285-1317,1999
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for universal prevention of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2022 Feb 10;2(2):CD013443. doi: 10.1002/14651858.CD013443.pub2. PMID 35141873